CLINICAL TRIAL: NCT04800783
Title: Development and Assessment of a New Ultrasound Score to Diagnose Swallowing Disorders in at Risk-out-patients
Brief Title: Diagnostic Accuracy of Aerodigestive Ultrasound for Predicting Swallowing Disorders
Acronym: DARC-VADOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Forcilles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02942-37
Record Dates: First submitted 2021-03-02; First posted 2021-03-16 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-03

CONDITIONS: Deglutition Disorders
Keywords: Swallowing disorders; Ultrasonography; Outpatients; Laryngeal; Tongue; Validation study
MeSH Terms: conditions — Deglutition Disorders; Laryngeal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective interventional study including consecutive patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swallowing disorders cohort (Other): All included patients will undergo an ultrasound assessment of the oral and laryngeal structures involved in the swallowing process.
  Interventions: Diagnostic Test: Swallowing ultrasound

INTERVENTIONS:
Diagnostic Test: Swallowing ultrasound — Ultrasound assessment of the tongue movement and thickening, the geniohyoid and suprahyoid muscles echogenicity, thickness and thickening, the hyoid bone elevation, and the number of swallowing trial.

SUMMARY:
Swallowing disorders management requires an accurate recognition of implicated anatomical structures and pathways. The usual clinical assessment of swallowing disorders lacks reliability and accuracy. The gold standard remains the videofluoroscopy. However, this imaging technique lacks reliability and standardisation. Moreover, videofluoroscopy is not easily available, time and material consuming and exposes patients to ionisation. Ultrasound imaging, which can be performed at the patient's bedside, is a non-invasive tool. It allows the evaluation of the main structures involved in all the swallowing pathways and may be a promising tool to assess the swallowing disorders. An ultrasound predictive model has never been developed to diagnose swallowing disorders.

The investigators aim to develop an ultrasound predictive model to diagnose swallowing disorders, and assess its reliability and accuracy.

One hundred outpatients at risk of swallowing disorders (neck cancer, neurological diseases, previous ICU stay) will be enrolled in the Dysphagia Diagnostic Unit at the Forcilles' Hospital, during a 2-year period.

All patients will undergo a clinical examination by a speech-language therapist, and a videofluoroscopy imaging in order to diagnose swallowing disorders. Then, an ultrasound examination will be performed by the ultrasonographer. The ultrasonographer will be blinded from the patient's status and previous clinical and imaging assessments. Severity of the swallowing disorder will be assessed by the Dysphagia Outcome and Severity Scale.

The tongue kinetics and thickness, the laryngeal movement and the suprahyoid muscles thickness and echogenicity will be assessed by ultrasonography.

Inter- and intra-reliability of ultrasound examination will be calculated. The threshold of each ultrasound measurement allowing the swallowing disorders will be estimated using the ROC curve analysis. Sensitivity and specificity of each ultrasound measurement will be estimated. A global ultrasound predictive model will be developed after selecting variables in logistic multivariable regression. Diagnostic accuracy of the global predictive model will also be assessed.

The investigators hope a high reliability and accuracy of the ultrasound predictive model in the swallowing disorders diagnostic. As ultrasonography is easy-to-perform, rapidly available, non-invasive and inexpensive, it may be a valuable alternative to videofluoroscopy in swallowing disorder diagnostic.

DETAILED DESCRIPTION:
Swallowing disorders management requires an accurate recognition of implicated anatomical structures and pathways. The usual clinical assessment of swallowing disorders lack of reliability and accuracy. The gold standard remains the videofluoroscopy. However, this imaging technique lacks reliability and standardisation. Moreover, videofluoroscopy not easily available is time and material consuming and implies ionisation. Ultrasound imaging, which can be performed at the patient's bedside, is a non-invasive tool. It allows the evaluation of the main structures involved in all the swallowing pathways and may be a promising tool for swallowing disorders assessment.

The investigators aim to develop an ultrasound predictive model to diagnose swallowing disorders, and assess its reliability and accuracy.

The investigators hope a high reliability and accuracy of the ultrasound predictive model in the swallowing disorders diagnostic. As ultrasonography is easy-to-perform, rapidly available, non-invasive and inexpensive, it may be a valuable alternative to videofluoroscopy in swallowing disorders diagnostic.

1. Hypothesis The investigators hypothesise that a new ultrasound predictive model is valid and reliable to diagnose swallowing disorder.
2. Objectives

   Primary objective:

   • To create a new ultrasound predictive model based on the most relevant ultrasound measurements of the swallowing structures.

   Secondary objectives:
   * To assess the accuracy of the ultrasound predictive model in the swallowing disorders diagnostic;
   * To assess the inter- and intra-reliability of the ultrasound measurements;
   * To assess the accuracy of each ultrasound measurements.
3. Study design:

   The prospective observational single-centre study will be performed per the ethical standards of the Declaration of Helsinki and will be reported according to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement.
4. Population:

   One hundred outpatients at risk of swallowing disorders (neck cancer, neurological diseases, previous ICU stay) will be enrolled in the Dysphagia Diagnostic Unit at the Forcilles' Hospital, during a 2-year period. All consecutive patients will be screened at hospital admission, and will be included if they satisfy the eligibility criteria. All patients will provide oral consent to participate, in accordance with the clinical research French laws. Duration of the patient's participation will take 3 hours.
5. Data collection Data will be recorded using a local case report form. Demographic data, comorbidities, medical and surgical history, reason for swallowing assessment will be recorded at inclusion. Clinical, videofluoroscopy and ultrasound measurements will also be recorded. On-site monitoring is planned every month.

   Participants will first undergo an ultrasound examination, then the clinical examination and videofluoroscopy imaging.
6. Ultrasound examination:

   Ultrasonography will be performed using a Sonosite E2 Expert ultrasound device (Digital Color Doppler Ultrasound System; Sonoscape medical corp. China) with a 7-10 MHz linear and a 3-5 MHz probes. Detailed information for ultrasound procedure is described in the research protocol. Ultrasonography will be performed with the patients in near-to-supine position (30°).

   The hyoid bone movement, tongue kinetics and geniohyoid muscle measurement will be performed in a sagittal plane with the curvilinear probe. The probe will be placed between the posterior border of the symphysis and the anterior margin of the hyoid bone.

   The anterior belly of digastric and geniohyoid muscles evaluation will be performed in a frontal plane with the linear probe. The probe will be placed in the submandibular area, behind the symphysis.

   Ultrasonographer will be blinded from all patients' status and previous examination. Reliability will be assessed in the first twenty participants. All ultrasound measurements will be repeated twice by the first ultrasonographer to assess the intra-operator reliability. A second ultrasound operator will perform all the ultrasound measurement, allowing the inter-operator reliability evaluation.
7. Videofluoroscopy (VFSS):

   VFSS is a radiographic procedure that provides a direct, dynamic view of oral, pharyngeal, and upper oesophageal function during swallowing. The radiologist and SLP work as a team to follow a standard protocol for conducting this examination.

   During this procedure, the speech-language therapist presents food and fluid mixed with barium. The barium is necessary to view structures via videofluoroscopy during the swallow. The following procedure will be followed: 5 ml of thin fluid; 5 ml of ultra-thick liquid; 5 ml of solid aliment, then 30 ml of thin fluid.

   The VFSS allow the assessment of the characteristics of the swallow and the patterns of bolus movement, including initiation of the swallow, nasopharyngeal reflux, pharyngeal clearance, and laryngeal penetration and aspiration.

   At any time, the radiologist may not initiate or stop the examination if it may be harmful to the patient. The reason to stop the test will be recorded.

   In case of penetration or aspiration, the speech language therapist will use the 'Penetration-Aspiration Scale'.
8. Statistical plan:

   Continuous variables will be expressed as the mean (± standard deviation) and compared using the Student's t test if the null hypothesis is not rejected by the Shapiro-Wilk test. Continuous variables will be expressed as the median (interquartile range) and compared with the Mann-Whitney U or Kruskal-Wallis test if the null hypothesis is rejected by the Shapiro-Wilk test. For categorical variables, the proportions of patients in each category will be calculated. Then the groups will be compared using Chi squared test.

   Continuous ultrasound variables will be dichotomised or grouped by class, depending on the linear relation between the logit of the swallowing disorder diagnostic and the ultrasound variable. The threshold for continuous ultrasound variables will be calculated with the ROC curve analysis.

   A multivariate logistic regression model will be carried out to assess the relation between swallowing disorders and ultrasound measures associated in univariate analyses. All statistically significant ultrasound variables will be included in the model. Variable selection will be stepwise, based on Akaike Information Criterion. To check multicollinearity between independent variables, the variance inflation factor will be calculated before performing multivariate logistic regression. Multicollinearity will be regarded as present when the variance inflation factor is > 5. Goodness of fit will be assessed by Hosmer-Lemeshow method.

   The outcome of each ultrasound variable from the multivariable logistic regression will be used to weight it in the global ultrasound predictive model.

   Intra- and inter-operator reliability will be assessed using the kappa coefficient for categorical variables or intra-class coefficients for continuous variables.

   For all tests, a p-value ≤ 0.05 will be considered statistically significant. All statistical analysis will be made using R software (version 3.6.1, www.R-project.org).
9. Sample size calculation:

The investigators based the sample size calculation on the number of independent variables which will be included in the logistic multivariable regression model. The investigators use the criterion of one variable per 10 events for binary logistic regression analysis. The investigators plan to include the 5 most relevant ultrasound measures in the model. As prevalence of swallowing disorders in our unit is estimated at 0.5, the investigators plan a sample size of 100 patients.

Reliability will be assessed on the first 20 patients. With an 80% predicted kappa, a minimal value of the kappa of 50%, 2 observations, a 95% certainty and a 80% power, 20 patients will be required.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients refered to swallowing assessment at the Forcilles' hospital;
* Medical indication to perform a videofluoroscopy;
* Ultrasonographer available;
* Age > 18 years old;
* Membership of a social insurance sheme;
* Patient provides consent.

Exclusion Criteria:

* Previous laryngectomy surgery;
* Refusal to participate in the study;
* Known pregnancy;
* Person subject to judicial health protection;
* Cognitive disorder incompatible with the understanding of instructions;
* Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Swallowing ultrasound predictive model development | Through study completion, an average of 2 years
  Selection of the most contributive ultrasound measures in the swallowing disorders diagnostic predictive model.

SECONDARY OUTCOMES:
Accuracy and reliability of ultrasound measure of hyoid bone movement | Through study completion, an average of 2 years
  Hyoid bone displacement will be recorded during swallowing. The video clips will be recorded in an external hard drive and then analyzed. The resting position of the hyoid bone will be used as axis coordinate system. The distance between resting position and during swallowing highlights the hyoid bone displacement. The hyoid bone displacement in x (anterior displacement) and y (superior displacement) axis will be measured in centimeters.
Accuracy and reliability of ultrasound measure of the tongue kinetics | Through study completion, an average of 2 years
  M-mode will be used to measure the vertical movement of the tongue (distance, in centimeters). The ultrasound line represents the tongue surface. The signal amplitude allows the assessment of vertical distance between the ultrasound line in resting position and during the swallowing.
  The time between the start of the movement and the back to the resting position will be assessed.
Accuracy and reliability of ultrasound measure of the digastric muscles | Through study completion, an average of 2 years
  Linear transducer will be used to obtain a coronal plane of suprahyoid muscles: anterior belly of digastrics muscle. The muscles activity during swallowing will be recorded. The frames will be frozed allowing the measure of the muscle thickness and Cross Sectional Area (CSA) of anterior belly of digastrics muscle. Thickness will be measured with calipers. To CSA quantification, a region of interest will be delimitated using free mode calipers. The CSA image will be used to quantity the echogenecity (grey level) with Image J software.
Accuracy and reliability of ultrasound assessment of the geniohyoid muscle | Through study completion, an average of 2 years
  Two different methods will be used: M-mode and B-mode. M-mode will be used to quantify the geniohyoid thickness at resting position and during swallowing. The ultrasound line represents geniohyoid muscle surface. The signal amplitude allows the assessment of muscle thickness.
  With B-mode method, the geniohyoid muscle thickness at resting position and during swallowing will be measured. The thickness will be measured in centimeters.
Inter and intra-operator reliability assessment of the swallowing ultrasound assessment | Through tweenty first inclusion completion, an average of 15 weeks
  Two operators will repeat the previous described outcomes measurement three times.
  The second ultrasound operator will perform all sonographic measurements following the first operator. Both ultrasound operators will be blinded from the patient's information. The second ultrasound operators will be blinded from the first ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Diaz Lopez, PT, Principal Investigator — Hôpital Forcilles-Fondation Cognacq-Jay
Locations (1):
- Hôpital Forcilles, Férolles-Attilly, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlie results in a publication will be uploaded in a repository platform.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data requesters must provide supporting documentation (e.g: research proposals) to the principal investigator. Request will be reviewed by the research committee of the sponsor.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04800783/Prot_SAP_ICF_002.pdf